CLINICAL TRIAL: NCT00147212
Title: A Phase II Study of Three Hour, Weekly Infusion of ET 743 (Yondelis) in Men With Advanced Prostate Cancer
Brief Title: ET 743 (Yondelis) in Men With Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); PharmaMar (Industry)
Responsible Party: Principal Investigator, Dror Michaelson, MD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-061
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2012-12

CONDITIONS: Prostate Cancer
Keywords: Advanced Prostate Cancer; Prostate Cancer; Trabectedin; ET 743; Yondelis
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): ET-743
  Interventions: Drug: ET 743

INTERVENTIONS:
Drug: ET 743 — ET-743 administered IV by 24-hr infusion every 3 weeks
  Other Names: Trabectedin; Yondelis

SUMMARY:
The main purpose of this study is to find out what effects (good or bad) trabectedin (ET743) has on men with advanced prostate carcinoma.

DETAILED DESCRIPTION:
* Treatment with trabectedin will be given once a week for three consecutive weeks with one week of no treatment. This four week period constitutes one cycle.
* Trabectedin is given as an infusion through a central venous catheter and is administered over 3 hours.
* On day 1 of each cycle a history, physical exam and blood tests will be performed and trabectedin will be administered.
* On day 8 and day 15 of each cycle blood work will be performed and trabectedin will be administered.
* Patients will continue to receive trabectedin as long as there is no disease progression or unacceptable side effects.
* Scans (CT, MRI or bone) or x-rays may be done while the patient is on the trial at the discretion of the physician.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Radiographically documented metastatic disease
* Surgical or chemical castration
* Prostate specific antigen (PSA) > 5 ng/ml
* Castration resistant prostate cancer (CRPC)
* One previous taxane-based chemotherapy regimen
* Eastern Cooperative Group (ECOG) performance status 0,1 or 2
* Neutrophil count > 1,500/ul
* Platelet count > 100,000/ul
* Serum bilirubin < 1.0 x upper limit normal (ULN)
* Serum alkaline phosphatase < 1.5 x ULN
* Asparate aminotransferase/Alanine aminotransferase < 2.5 x ULN
* Albumin > 2.5 g/dl
* Serum creatinine < 1.5 x ULN
* Prior hormonal therapy

Exclusion Criteria:

* Chemotherapy treatment within 4 weeks of study entry
* Patient not employing adequate contraception
* Serious illness or medical conditions, specifically: uncontrolled congestive heart failure or history of myocardial infection or active angina pectoris within 6 months; active infectious process; chronic active liver disease, including chronic hepatitis B, C or cirrhosis
* Current anti-cancer treatment with any non-FDA approved investigational drug

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dror Michaelson, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Masachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Completed
Groups:
- Trabectedin: Experimental arm treated with trabectedin (ET-743)
Period: Overall Study
Arm/Group | Trabectedin
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Trabectedin
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 65 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 50
Region of Enrollment [Number; unit: participants]
  Spain | 4
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: The Number of Men With Advanced Prostate Cancer Treated With Trabectedin Who Have a PSA Response
Description: Prostate specific antigen (PSA) response rate, as defined by the PSA Working Group Criteria (see Bubley et al, J Clin Oncol. 1999 Nov;17(11):3461-7)
Time Frame: Participants were followed until disease progression, an average of 6 months
Population: Intent to treat
Measure: Number; unit: participants
Groups:
- Trabectedin: Men with metastatic castration resistant prostate cancer (CRPC) treated with trabectedin
Arm/Group | Trabectedin
Number analyzed (Participants) | 50
participants | 7 [0 to 50]

ADVERSE EVENTS:
Arm/Group | Trabectedin
Serious Adverse Events (participants affected / at risk) | 10/50
Other Adverse Events (participants affected / at risk) | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trabectedin (N=50)
Neutropenia (Blood and lymphatic system disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No